CLINICAL TRIAL: NCT02595021
Title: A Phase II Study of Total or Subtotal Colectomy in Stage IIIC and Stage IV Epithelial Ovarian, Fallopian Tube, and Primary Peritoneal Cancer (EOC, FTC, PPC)
Brief Title: Total/Subtotal Colectomy in Ovarian Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Gynecologic Oncology Group (Other Government)
Collaborators: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: zsfud-obgyn-004
Record Dates: First submitted 2015-09-18; First posted 2015-11-03 (Estimated); Last update posted 2016-07-26 (Estimated); Status verified 2016-07

CONDITIONS: Epithelial Ovarian Cancer; Fallopian Tube Cancer; Primary Peritoneal Carcinoma; Secondary Malignant Neoplasm of Large Intestine
Keywords: Total or subtotal colectomy; Ovarian cancer; Complications; One-year disease-free survival; Stage IIIc; Stage IV
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial; Fallopian Tube Neoplasms; Ovarian Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Total or Subtotal Colectomy (Experimental): all patients who underwent total colectomy(removal of the large intestine from ileum to the rectum. After it is removed, the end of the small intestine is sewn to the rectum) or subtotal colectomy(removal of transverse colon, descending colon, sigmoid colon to the rectum. After it is removed, the end of the ascending colon is sewn to the rectum)as part of optimal cytoreductive surgery
  Interventions: Procedure: Total or Subtotal Colectomy
- Other Bowel Resection (Active Comparator): all patients who underwent partial intestinal resection as part of optimal cytoreductive surgery
  Interventions: Procedure: Other Bowel Resection

INTERVENTIONS:
Procedure: Total or Subtotal Colectomy — Resect all or most parts of the colon: with total or subtotal colectomy as a part of optimal cytoreductive surgery(residual disease <=0.5cm)
  Other Names: Radical surgery; Total Colectomy; Subtotal Colectomy
  Arms: Total or Subtotal Colectomy
Procedure: Other Bowel Resection — Resect part of the colon or small intestine: with other types of bowel resection as a part of optimal cytoreductive surgery(residual disease <=0.5cm)
  Other Names: Partial Colectomy; Small bowel resection
  Arms: Other Bowel Resection

SUMMARY:
The purpose of this study is to evaluate the safety and one year disease-free survival of total or subtotal colectomy and proctocolectomy in stage IIIc and stage IV epithelial ovarian, fallopian tube, and primary peritoneal cancer (EOC, FTC, PPC).

DETAILED DESCRIPTION:
This trial is to assess the perioperative complications, hospitalization expenses and days, and one year disease-free survival of patients who underwent total or subtotal colectomy as part of the surgical procedures for ovarian cancer, versus partial intestinal resection in the therapy for ovarian cancer.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years and ≤ 75 years.
* Epithelial ovarian cancer, fallopian tube cancer, primary peritoneal carcinoma with pathology confirmed International Federation of Gynecology and Obstetrics (FIGO) stage IIIc or IV
* Extensive colonic metastasis, tumor involving the major part of bowel surface and/or mesentery
* Optimal cytoreductive surgery, including hysterectomy, bilateral salpinges-oophorectomy, omentectomy, and resection of all metastatic lesions, with a residual disease no more than 0.5cm
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2.
* American Society of Anesthesiologists (ASA) performance 1-2.
* Follow-up available.
* Written informed consent.

Exclusion Criteria:

* Low-malignant potential ovarian tumor.
* Patient who underwent enterostomy in the surgery procedure.
* Tumor involving small intestine alone.
* More than 2 anastomoses.
* Other condition that could interfere with provision of informed consent, compliance to study procedures, or follow-up.
* Prior invasive malignancies within the last 5 years showing activity of disease.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2015-07; Primary Completion 2017-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Postoperative complications | up to 30 days after surgery
  Assessed by Common Terminology Criteria for Adverse Events version 4.0 up to 30 days after surgery

SECONDARY OUTCOMES:
The rate of 12- month- disease non-progression | up to 12 months
  Number of patients without progression in 12 months (From date of first chemotherapy until the date of first documented progression, assessed up to 12 months)
Initiation of the first cycle chemotherapy | up to 12 weeks
  To compare the date between surgery and initiation of the first cycle chemo
Hospitalization expenses | up to 12 weeks
  the cost during hospital stay
Hospitalization days | up to 12 weeks
  length of hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Rongyu Zang, MD,PhD, Principal Investigator — Shanghai Zhongshan Hospital
Locations (1):
- Fudan University Shanghai Zhongshan Hospital, Shanghai, Shanghai Municipality, China

REFERENCES:
- See also: Shanghai Gynecologic Oncology Group — http://www.ShanghaiGOG.org